CLINICAL TRIAL: NCT04036214
Title: Selective Laser Trabeculoplasty (SLT): Efficacy and Safety Outcomes of Optometrist (OD) Performed SLT
Brief Title: Efficacy and Safety Outcomes of Optometrist Performed Selective Laser Trabeculoplasty (SLT)
Acronym: SLT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northeastern State University (Other)
Responsible Party: Sponsor
Other Study IDs: NSUOCO0001
Record Dates: First submitted 2019-07-17; First posted 2019-07-29 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Primary Open-Angle Glaucoma, Unspecified Eye; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Selective Laser Trabeculoplasty — Selective Laser Trabeculoplasty Laser

SUMMARY:
To measure the efficacy and safety outcomes of SLT performed by optometrists.

DETAILED DESCRIPTION:
Participants will undergo a pre-procedure examination in order to record baseline findings and to determine if they meet the inclusion criteria in order to undergo the procedure. Participants will undergo the SLT procedure and will be examined at 1 hour, 1 week and 6 weeks. Follow up examinations will evaluate eye pressure reduction and post-procedure complications. The rate complication post-procedure are typically low.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent;
2. At least 18 years of age, male or female, of Native American or Alaskan Native descent;
3. Diagnosed with primary open angle glaucoma or ocular hypertension;
4. Documented intraocular pressure greater than or equal to 23 mmHg;
5. No prior glaucoma treatment unless treated with one topical drop.

Exclusion Criteria:

1. History of trauma or ocular surgery within the last 6 months;
2. History of corneal dystrophy;
3. Current use of topical or systemic steroids;
4. Advanced or severe glaucomatous findings based on comprehensive examination;
5. Diagnosed with other types of glaucoma such as pseudoexfoliation syndrome, pigmentary glaucoma, normal tension glaucoma, and other additional glaucoma subtypes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing patients at primary eye care optometric facilities.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure via Goldmann tonometry | 6 weeks
  Pre and Post Procedure Intraocular Pressure will be measured using a Goldmann tonometer and will be measured in millimeters of Mercury (mmHg). Percent change in intraocular pressure will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Nate Lighthizer, OD, Principal Investigator — Northeastern State University
Locations (1):
- Northeastern State University, Tahlequah, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No